CLINICAL TRIAL: NCT02941289
Title: Visuospatial Attention and Eye Movement Behaviour in Patients With Alzheimer's Disease When Searching in Realistic Scenes and a Natural Setting: Exploring Perceptual and Cognitive Mechanisms and Their Relationships With IADLs
Brief Title: Visuospatial Attention, Eye Movements and Instrumental Activities of Daily Living (IADLs) in Alzheimer's Disease
Acronym: ARVA-MA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-AOI-06
Record Dates: First submitted 2016-05-30; First posted 2016-10-21 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alzheimer's patient (Experimental): Probable diagnosis of Alzheimer's disease with a mild impairment (MMSE 20-26) according to DSM IV diagnosis criteria
  Interventions: Procedure: visual search performance of everyday objects in realistic scenes
- Control patient (Active Comparator): patient with MMSE score equal or > 27
  Interventions: Procedure: visual search performance of everyday objects in realistic scenes

INTERVENTIONS:
Procedure: visual search performance of everyday objects in realistic scenes

SUMMARY:
The aim is to understand which components of attentional deployment and selection are impaired in AD during searching in realistic scenes on a computer screen (Experiment 1) and in a natural setting (Experiment 2).The investigators will also examine how deficits in visual exploration may be related to impairments in semantic, long-term memory (LTM) and working memory (WM) representations by manipulating the semantic consistency between the target and its visual surroundings, and the type of target cue (abstract vs. precise), respectively. Perceptual saliency of target and distractor objects will be also manipulated in Expt.1, In Expt.2, in order to determine how deficits in visual exploration may be involved in the IADL deficits shown by AD patients, participants at each trial will be required to search in a natural settings different types of targets and then to perform an IADL using five objects, among which one of the searched targets. Measures analysed: for the search tasks (Expt. 1 and 2): eye movements in different search phases, accuracy and response times; for IADLs tasks (Expt. 2): eye movements during action planning and execution, motor efficiency (number and types of action performed), time to terminate the activity. Compared to controls, the investigators expect that AD patients will have reduced ability using scene semantic LTM in order to locate the objects, greater attentional capture from highly salient features and greater search performance impairment when higher WM resources are required (abstract target cues). The investigators also expect that their performance at IADLs will be less efficient and, in particular, less organized than control, with reduced advantage of eye guidance.

DETAILED DESCRIPTION:
It has been well established that visual attention declines early in Alzheimer's Disease (AD). Little is known about visual search in AD, in particular in relation with functional autonomy. The crucial role of the parietal cortex in visuospatial attention and instrumental activities of daily living (IADLs), and the presence of early parietal damage in AD suggest that IADLs may also be impaired early. The aim is to understand which components of attentional deployment and selection are specifically impaired in AD during searching in static realistic scenes presented on a computer screen (Experiment 1) and in a natural setting (Experiment 2: different regions of a room, furnished with different types of objects indicating different possible daily-living environments, like a kitchen or an office). More precisely, the investigators will examine how deficits in visual exploration during search for a target objects may be related to impairments in semantic, long-term memory (LTM) and in working memory (WM) representations by manipulating, respectively, semantic consistency between the target and type of its visual surrounding (scene context, in Expt. 1, or type of co-occurring objects, in Expt 2).and the type of prior information supplied about the target object (abstract - i.e., verbal - or precise, - i.e., pictorial), In Expt. 1 the investigators will also manipulate the perceptual salience (low-level feature: luminance, colour, orientation, etc.) of the target and the distractor objects within the scene. Second, to determine how deficits in visual exploration during search for specific objects may be involved in the deficits of IADL in AD, the investigators will analyse search behaviour in the natural setting, requiring location of three different targets (semantically consistent/related to an IADL, semantically consistent/ non-related to an IADL, semantically inconsistent/non-related). The investigators will required participants to perform an IADL after each search (four trial in total) using, among other four objects, the IADL-related searched target). In Expt. 1 the investigators will test three groups of participants: the AD group (at early stage of the disease), a matched control group of healthy elderly people and a control group of young, healthy individuals. The investigators will examine search performance (accuracy and response time) and oculomotor behaviour during the different search phases (initiation, scene scanning, target verification). They expect that AD patients will have reduced search performance compared to both control groups, which will be also reflected by reduced oculomotor efficiency during the overall search process. Moreover, they hypothesize that patients will be less able to use semantic memory of the type of scene in order to locate the target (reduced benefit of scene consistency), will be strongly disadvantaged in case of higher WM load (abstract target cue) and, finally, will be more influence by perceptual, low-level factors (stronger effect of salience). In Exp. 2, they will test an AD group and a control group of healthy, matched, old controls. With respect to the search tasks, they will analyse the effect of target semantic consistency, target relatedness to IADL and type of target cue (abstract vs. precise). In doing so, they will consider search performance (accuracy and response times) and oculomotor behaviour during search in terms of order and number of object fixated, and duration of their fixation. With respect to the IADLs, they will analyse eye guidance on current action and efficiency of the whole IADL in terms of type and number of actions performed and time to perform the overall activity. They expect that the patterns of eye movements in AD patients will be similar during search and IADLs, with numerous intrusions of distractors and frequent reselections of the same objects. Moreover, they expect that their performance at IADLs will be less efficient than controls, in terms of both action speed and organisation. The use of a natural setting and the analysis of spontaneous oculomotor behavior of patients will improve the ecological validity of research on attentional deficits in AD. This study can also contribute to innovative solutions for diagnosis and treatment, and help research on subjective change in attention and visuospatial function in AD

ELIGIBILITY:
Inclusion Criteria: Control participants

* Male and female
* Age between 65 and 75 years old
* MMSE score equal or > 27
* Normal visual acuity (with or without correction to normality)
* Subjects with a score of 0 on " tremors " and " rigidity " items of UPDRS III scale
* Subjects without major depression criteria according to DSM IV-R
* No apathy according to diagnostic criteria of apathy
* Signed informed consent

Inclusion Criteria: Alzheimer's disease patients

* Male and female
* Age between 65 and 75 years old
* Probable diagnosis of Alzheimer's disease with a mild impairment (MMSE 20-26) according to DSM IV diagnosis criteria
* Normal visual acuity (with or without correction to normality)
* Subjects with a zero score on " tremors " and " rigidity " items of UPDRS III scale
* Signed informed consent

Exclusion Criteria:

* Controls with neurological and/or psychiatric pathologies
* AD patients with neurological and/or psychiatric pathologies unrelated to AD
* AD patients with vascular dementia suspicion in addition to the probable diagnosis of AD
* AD patients with MMSE score < 20
* Individuals with abnormal visual acuity (i.e., glaucoma, cataract sufficiently severe that limited vision…)
* Individuals with motor disorders, Parkinsonism…
* Receiving drug treatments that could alter cognitive functions

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Total number of fixations during search | at 2 weeks
  Oculomotor behavior and search performance in AD patients compared to elderly controls in a computerized visual search task using realistic scenes (Experiment 1), as well as when searching for specific objects in a real setting and during activities of daily living (Experiment 2).
Total duration of fixations during search | at 2 weeks
  This is the eye movement parameters that the investigators will analyze in the data

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramzaoui H, Faure S, David R, Spotorno S. Top-down and bottom-up sources of eye-movement guidance during realistic scene search in Alzheimer's disease. Neuropsychology. 2022 Oct;36(7):597-613. doi: 10.1037/neu0000797. Epub 2022 Jul 7. PMID 35797174
- [Derived] Ramzaoui H, Faure S, Spotorno S. Top-down and bottom-up guidance in normal aging during scene search. Psychol Aging. 2021 Jun;36(4):433-451. doi: 10.1037/pag0000485. PMID 34124920